CLINICAL TRIAL: NCT04729556
Title: Safety Evaluation of a Film-forming Cream Containing Sericin and Chitosan for Pressure Sore Treatment in Healthy Volunteers
Brief Title: Safety Evaluation of Sericin-chitosan Cream in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Pornanong Aramwit, Pharm.D., Ph.D, Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EC 19310-20
Record Dates: First submitted 2021-01-25; First posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Pressure Sore; Safety Issues
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sericin and chitosan cream (Experimental): A flim-forming cream containing sericin and chitosan cream. Apply sericin and chitosan cream on the back area of healthy volunteers and cover with self-adhesive nonwoven fabric in induction phase I (72 hours), induction phase II (72 hours), and challenge phase (72 hours).
  Interventions: Device: Sericin and chitosan cream
- Cavilon (Active Comparator): Active control is a commercial cream containing dimethicone as the substance forms a durable, thin, and transparent film. The cream is used as a moisturizer to prevent the skin against irritation, dryness, and pressure ulcers.
  Apply sericin and chitosan cream on the back area of healthy volunteers and cover with self-adhesive nonwoven fabric in induction phase I (72 hours), induction phase II (72 hours), and challenge phase (72 hours).
  Interventions: Device: Sericin and chitosan cream

INTERVENTIONS:
Device: Sericin and chitosan cream — A novel film-forming cream containing sericin and chitosan

SUMMARY:
A prospective, randomized, active-controlled clinical trial was conducted to evaluate safety of sericin-chitosan cream in healthy volunteers.

DETAILED DESCRIPTION:
A prospective, randomized, active-controlled clinical trial was conducted to initially evaluate safety of sericin-chitosan cream in comparison with a commercially available cream containing dimethicone for pressure sore treatment in healthy volunteers. The results of this study provided preliminary safety profile of sericin-chitosan cream before conducting the further clinical trial in specific population (pateints with early-stage pressure sore).

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers at the age of 20 - 65 years
* voluntarily sign inform consent

Exclusion Criteria:

* Diagnosed with chronic skin conditions (e g. eczema and psoriasis) and immunocompromised diseases
* Allergic to silk sericin and chitosan, and dimethicone
* Received immunosuppressive therapy, antihistamine, and corticosteroid drugs two weeks before study enrollment.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
Skin erythema index | 17 days
  Erythema index will be measured using Cutometer (Mexameter). There is no unit. Higher value mean higher risk of post inflammatory reaction.
Skin melanin index | 17 days
  Melanin index will be measured using Cutometer (Mexameter). There is no unit. Higher value mean higher risk of post inflammatory reaction.

SECONDARY OUTCOMES:
Visual skin irritation | 17 days
  Photographs of the contact skin area will be used for evaluating the presences and severity of skin irritation (rash, edema, papules, vesicles, and bullae) by dermatologists.
Self-report topical side effects: rash, edema, vesicles, and itching | 17 days
  Participants will be asked to self-monitor topical side effects: rash, edema, vesicles, and itching (if any), and then inform the investigators.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pharmacy Practice, Faculty of Pharmaceutical Sciences, Chulalongkorn Unviersity, Bangkok, Thailand